CLINICAL TRIAL: NCT05798754
Title: Correlation of Standard Loss of Resistance Technique Versus the CompuFlo®-Assisted Technology for Thoracic Epidural Space Identification
Brief Title: Efficacy of CompuFlo® Technology in Thoracic Epidural Space Identification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General and Maternity Hospital of Athens Elena Venizelou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21/03/2023/ID
Record Dates: First submitted 2023-03-21; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Thoracic Epidural Space Identification
Keywords: thoracic; epidural space; loss of resistance technique; CompuFlo® technology
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Prospective blind, non-inferiority randomized trial
Who Masked: Outcomes Assessor
Masking Description: Member of the study group that assesses the epidural's success
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group LOR (Active Comparator): The thoracic epidural space will be identified by the loss of resistance technique.
  Interventions: Procedure: Loss of resistance (LOR) technique
- Group C (Active Comparator): The thoracic epidural space will be identified by the CompuFlo® technology.
  Interventions: Device: CompuFlo® technology

INTERVENTIONS:
Procedure: Loss of resistance (LOR) technique — The thoracic epidural space will be identified by the loss of resistance (LOR) technique
  Arms: Group LOR
Device: CompuFlo® technology — The thoracic epidural space will be identified by the CompuFlo® technology
  Arms: Group C

SUMMARY:
The aim of this non inferiority trial is to assess the efficacy of CompuFlo® technology to identify the thoracic epidural space in relation to the gold standard loss of resistance technique.

DETAILED DESCRIPTION:
This non inferiority trial shouts to adress whether the CompuFlo® technology to identify the thoracic epidural space is less efficacious to the gold standard loss of resistance technique (LOR). After informed signed consent patients that will be subjected to gynecological operations and meet the inclusion criteria will be eligible to participate. All operations will be performed under general anesthesia and thoracic epidural analgesia regardless of study arm. Patients will be randomly allocated into two study groups. In the first study group (Group LOR) the thoracic epidural space will be identified by the LOR technique and in the second study group (Group C) by the CompuFlo® technology. The primary outcome is the percentage of thoracic epidural space identification success in either study group.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) Physical Status Classification System I-III Body mass index: 18 -35 kg/m2 Gynecological laparotomy with midline incision under general anesthesia and thoracic epidural analgesia

Exclusion Criteria:

Patients' denial to participate in the study ASA Physical Status Classification System >IV Contraindications to epidural analgesia Patients with sepsis Patients with pre-existing neurologic deficits Pre-existing operations in the thoracic spinal cord Emergency operations Patients with end-stage cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of successful thoracic epidural space identification | Loss of sensation to cold 20 min after the first dose administered through the epidural catheter
  The success of the thoracic epidural space identification

SECONDARY OUTCOMES:
Percentage of successful thoracic epidural space identification by the first attempt | Loss of sensation to cold 20 min after the first dose administered through the epidural catheter during the first attempt
  Percentage of successful thoracic epidural space identification by the first attempt
Number of attempts to successful thoracic epidural space identification | Number of attempts to successful thoracic epidural space identification up to a maximum of 3 adressed as loss of sensation to cold 20 min after the first dose administered through the epidural catheter
  Number of attempts to successful thoracic epidural space identification
Time to identify the thoracic epidural space | Time to insertion of epidural needle (Tuohy) in the supraspinous ligament to insertion of the epidural catheter
  Time to identify the thoracic epidural space
Adverse events | From epidural needle insertion up to 72 hours postoperatively
  Adverse events (dural puncture, epidural hematoma, neurological deficit)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Stroumpoulis, PhD, Study Director — General and Maternity Hopsital of Athens Helena Venizelou
Locations (1):
- "Elena Venizelou" General and Maternity Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No